CLINICAL TRIAL: NCT05133765
Title: Optimising Glycaemia Around Dynamic Physical Exercise With Advanced Hybrid-closed-loop Therapy Use in Type 1 Diabetes: ''The SMART Study''
Brief Title: The SMART B Exercise Study :''The SMART Study''
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Swansea University (Other)
Responsible Party: Principal Investigator, Merete Bechmann Christensen, Principal Investigator, MD, PhD, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SMART B
Record Dates: First submitted 2021-09-14; First posted 2021-11-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Insulin Infusion Systems

STUDY DESIGN:
Intervention Model Description: Three period randomised cross-over clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMART B1 - Usual care insulin pump (Experimental): Usual care pump therapy arm with carbohydrate consumption before exercise
  Interventions: Device: Insulin pump
- SMART B2 - Advanced hybrid closed loop insulin pump with carbohydrates before exercise (Experimental): Advanced hybrid closed loop therapy arm with carbohydrate consumption before exercise
  Interventions: Device: Insulin pump
- SMART B3 - Advanced hybrid closed loop insulin pump with carbohydrates during exercise (Experimental): Advanced hybrid closed loop therapy arm with carbohydrate consumption during exercise
  Interventions: Device: Insulin pump

INTERVENTIONS:
Device: Insulin pump — Alterations in insulin pump therapy or carbohydrate consumption

SUMMARY:
Despite the established health benefits conveyed by physical activity for people with type 1 diabetes (T1D), participation rates remain low, with fear of hypoglycaemia, lack of freedom to engage in unplanned activities, and uncertainty in making appropriate adjustments to insulin and nutritional therapy reported as the leading barriers to regular exercise engagement. Indeed, the synergistic glucose lowering effects of peripheral hyperinsulinaemia and exercising muscle tissue accentuate the risk of exercise-related hypoglycaemia for individuals with T1D, particularly if performed post-prandially. Hence, the introduction of commercially available artificial pancreas systems, also known as ''advanced hybrid-closed-loop'' (AHCL) systems, that regulate insulin rates with minimal user interaction constitute compelling therapeutic aids with clinically relevant potential. Nevertheless, we know little about their safe and efficacious integration around dynamic physical exercise. Nor do we know how alterations in carbohydrate fueling strategies around exercise effect subsequent glucose trends.

This study aims to 1) compare the efficacy of an AHCL system versus usual care insulin pump therapy, with carbohydrates taken before or during exercise, in optimising TIR around dynamic physical exercise and 2) explore the influence of carbohydrate intake before versus during exercise on the metabolomic, hormonal and physiological responses to exercise.

DETAILED DESCRIPTION:
Following successful completion of a screening visit, participants will attend the laboratory to complete 3 experimental visits during which they will undertake a 45-minute bout of moderate intensity continuous exercise on a bicycle ergometer at ~60% of the individualised VȮ2max. Prior to commencing exercise, participants will consume a standardised low-glycaemic index, carbohydrate-based meal (equating to 0.75g.CHO.kg.bm-1) with, or without, a 25% reduction in their meal-time insulin dose as well as with carbohydrates before or during exercise (according to the randomisation). Venous blood glucose sampling will be taken in 15-minute intervals leading into and after exercise with 5-minute intervals performed during exercise. Samples will be used to retrospectively cross-compare the metabolic, hormonal, and physiological responses between visits. Visits 1 & 2 will be separated by ≥14 days to ensure adequate familiarisation with the AHCL system whilst visits 2 & 3 will be separated by ≥3days. Each participant will undertake 1 screening and 3 experimental visits equating to a total of 80 study visits.

ELIGIBILITY:
Inclusion Criteria:

* • Type 1 diabetes ≥2 years.

  * HbA1c;

    * 58-63 mmol/mol (maximum 30% of participants) OR
    * ≥ 64 mmol/mol (minimum 70% of participants)
  * Insulin pump treatment ≥12 months
  * CGM or isCGM use ≥6 months
  * Novorapid use ≥4 weeks
  * Carbohydrate counting and use of the insulin pump bolus calculator for most snacks and meals.
  * Carbohydrate intake >80 grams per day (assessed by review of intake recorded in the insulin pump during the 2 weeks prior to the screening visit)

Exclusion Criteria:

* • Breast-feeding, pregnancy or planning to become pregnant.

  * Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start.
  * Use of hybrid closed-loop systems
  * Daily use of paracetamol (acetaminophen)
  * Alcohol or drug abuse.
  * Severe cardiac disease or retinopathy contraindicating HbA1c <53 mmol/mol.
  * Other concomitant medical or psychological condition that according to the investigator's assessment makes the person unsuitable for study participation.
  * Lack of compliance with key study procedures at the discretion of the investigator.
  * Unacceptable adverse events at the discretion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Comparison of TIR in blood glucose values during, and 1-hour after, dynamic physical exercise | 0 minutes to +105 minutes
  Comparison of the amount of time spent with blood glucose values within the target range during, and 1-hour after, dynamic physical exercise

SECONDARY OUTCOMES:
To compare the influence of carbohydrate feeding before versus during exercise on the physiological responses to dynamic physical exercise | 0 minutes to +45 minutes
  To compare the influence of carbohydrate feeding before versus during exercise on the physiological responses to dynamic physical exercise

OTHER OUTCOMES:
Comparison of the maximum BG concentration | -90 minutes to +105 minutes
  Comparison of the maximum blood glucose concentration before, during and for 1 hour after physical exercise
Comparison of the minimum BG concentration | -90 minutes to +105 minutes
  Comparison of the minimum blood glucose concentration before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of standard deviation in BG concentrations | -90 min to +105 minutes
  Comparison of standard deviation in blood glucose concentrations before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of mean BG concentrations | -90 minutes to +105 minutes
  Comparison of mean blood glucose concentrations before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of the depth of BG hypoglycaemic events | -90 minutes to +105 minutes
  Comparison of the depth of blood glucose hypoglycaemic events before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of the occurrence of BG hypoglycaemic events | -90 minutes to +105 minutes
  Comparison of the occurrence of blood glucose hypoglycaemic events before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
ΔBGexercise: Comparison of the changes in BG during exercise | 0 minutes to +45 minutes
  ΔBGexercise: Comparison of the changes in blood glucose during exercise before, during physical exercise (i.e., 0 min to +45min)
ΔiGexercise: Comparison of the changes in iG during exercise | 0 minutes to +45 minutes
  ΔiGexercise: Comparison of the changes in interstitial glucose during exercise during physical exercise (i.e., 0 min to +45min)
ΔiGfeeding: Comparison of the changes in iG after feeding | -90 minutes to 0 minutes
  ΔiGfeeding: Comparison of the changes in interstitial glucose after feeding before physical exercise (i.e., -90 min to 0 min)
Comparison of TBR level 2 in iG values | -90 minutes to +105 minutes
  Comparison of the amount of time spent with interstitial glucose values below the target range level 2 before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of TBR level 1 in iG values | -90 minutes to +105 minutes
  Comparison of the amount of time spent with interstitial glucose values below the target range level 1 before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of TAR level 1 in iG values | -90 minutes to +105 minutes
  Comparison of the amount of time spent with interstitial glucose values above the target range level 1 before, during and for 1 hour after physical exercise (i.e., -0 min to +105min)
Comparison of TAR level 2 in iG values | -90 minutes to +105 minutes
  Comparison of the amount of time spent with interstitial glucose values after the target range level 2 before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of mean iG concentrations | -90 minutes to +105 minutes
  Comparison of mean interstitial glucose concentrations before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of the standard deviation in iG concentrations | -90 minutes to +105 minutes
  Comparison of the standard deviation in interstitial glucose concentrations before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of the coefficient of variation in iG concentrations | -90 minutes to +105 minutes
  Comparison of the coefficient of variation in interstitial glucose concentrations before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of the minimum iG concentration | -90 minutes to +105 minutes
  Comparison of the minimum interstitial glucose concentration before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)
Comparison of the maximum iG concentration | -90 minutes to +105 minutes
  Comparison of the maximum interstitial glucose concentration before, during and for 1 hour after physical exercise (i.e., -90 min to +105min)

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] McCarthy OM, Christensen MB, Kristensen KB, Schmidt S, Ranjan AG, Bain SC, Bracken RM, Norgaard K. Glycemia Around Exercise in Adults with Type 1 Diabetes Using Automated and Nonautomated Insulin Delivery Pumps: A Switch Pilot Trial. Diabetes Technol Ther. 2023 Apr;25(4):287-292. doi: 10.1089/dia.2022.0542. Epub 2023 Feb 16. PMID 36724311
- [Derived] McCarthy OM, Kristensen KB, Christensen MB, Schmidt S, Ranjan AG, Nicholas C, Bain SC, Norgaard K, Bracken R. Metabolic and physiological responses to graded exercise testing in individuals with type 1 diabetes using insulin pump therapy. Diabetes Obes Metab. 2023 Mar;25(3):878-888. doi: 10.1111/dom.14938. Epub 2023 Jan 3. PMID 36482870